CLINICAL TRIAL: NCT04842929
Title: Treatment of Depression in the Elderly With Repetitive Transcranial Magnetic Stimulation (rTMS) Using Theta-burst Stimulation (TBS): Randomized, Double-blind, Sham-controlled, Clinical Trial
Brief Title: Magnetic Randomized Trial in Elderly Depressed
Acronym: MrTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Leandro Valiengo, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2.643.551
Record Dates: First submitted 2021-01-20; First posted 2021-04-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; geriatric depression; repetitive transcranial magnetic stimulation (rTMS); theta-burst stimulation (TBS); elderly
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Stimulation (Active Comparator): Active Comparator: Active stimulation with pulses emitted according to intervention description
  Interventions: Device: Transcranial magnetic stimulation
- Sham Stimulation (Sham Comparator): Sham Comparator: The blinding will be done with a sham coil, which consists of a coil that reproduces the sound that the true coil does, but without generating the magnetic field.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — The coil will be positioned in the prefrontal dorsolateral cortex, with intermintent TBS (TBSi) mode on the left and continuous TBS (TBSc) on the right. 1800 pulses will be used on each side, totaling 10 minutes of total duration. There will be 20 consecutive sessions, one per day, except on weekends and holidays, totaling around 4 weeks. A day of stimulation with the same technique will be done in the 6th week, 8th week and 12th week.

SUMMARY:
Major depressive disorder (MDD) is a common psychiatric condition, mostly treated with antidepressant drugs, which are limited for issues such as refractoriness, adverse effects and drug interactions, especially in the elderly population. In this context, the investigators investigate a non-pharmacological treatment known as recurrent transcranial magnetic stimulation (rTMS) with the theta-burst stimulation (TBS) method for the treatment of geriatric depression. This treatment modality has almost no adverse effects and avoids the risk associated with polypharmacy, providing an interesting alternative to antidepressant treatments. Our aim is to evaluate TBS efficacy in the treatment of geriatric depression in a randomized, double-blind, placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Recurrent transcranial magnetic stimulation (rTMS) is a consolidated procedure for the treatment of depression, with several meta-analyzes demonstrating its efficacy. The theta-burst stimulation (TBS) method is a modification of the usual rTMS protocol. As a new protocol, there are still few studies evaluating its efficacy in treatment of major depression, although a recently published meta-analysis has pointed to benefits of this therapeutic modality. To date, there are no studies published with this method for the treatment of geriatric depression. This study will be a randomized, placebo-controlled, double-blind clinical trial to evaluate the efficacy of theta-burst rTMS in the treatment of major depressive disorder in the elderly, randomizing 108 subjects to the experimental (TBS) and comparative (sham) groups. The coil will be positioned in the dorsolateral prefrontal cortex, with intermittent TBS (iTBS, stimulatory) mode on the left and continuous TBS (cTBS, inhibitory) on the right. Stimulation protocol consists of 1800 pulses on each brain hemisphere, totaling a ten minutes session. There will be 20 consecutive sessions, one a day, except on weekends and holidays. The cycle of continuous intervention will last approximately four weeks, after which applications with the same technique will be performed at the end of weeks 6, 8 and 12. Clinical outcome measures will be obtained on eight occasions: treatment baseline, and after 1, 2, 4, 6, 8 and 12 weeks of onset. The main clinical outcome will be measured using the Hamilton Depression Scale (HDRS), comparing baseline scores with those obtained after 6 weeks of treatment. As secondary endpoints, we will use the Global Clinical Impression Scale (CGI), the CIRS (Cumulative Illness Rating Scale), the Geriatric Depression Scale (GDS), the intermediate scores obtained on the HDRS scale, the Positive and Negative Affect Scale (PANAS), the Montgomery-Asberg Depression Rating Scale (MADRS), and variations in serum BDNF concentrations; all these evaluation tools have validated versions in Portuguese. As tolerability and safety parameters, the incidence of adverse events and the occurrence of manic/hypomanic symptoms will be evaluated by the Young Mania Scale (YMRS). TBS stimulation will be evaluated in terms of safety, tolerability and effectiveness for the treatment of major depression in the elderly, possibly becoming another therapeutic option useful for patients with poor response or contraindications to the use of antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder;
* Patients older than 60 years
* Hamilton equal or higher than 17

Exclusion Criteria:

* Other mental disorders (alcohol or drug addiction, psychotic disorders, dementia, bipolar disorder);
* Presence of serious neurological or clinical diseases;
* Resence of severe suicidal ideation and CIRS (Cumulative Illness Rating Scale) score> 7, characterizing a set of clinical morbidities that could impair adherence to the research protocol, bipolar disorder and/or presence of manic symptoms (hypo) demonstrated with more than 8 points in the Young Mania Rating Scale.
* Metal implants;
* Epilepsy or electronics in the cephalic segment;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Changes in Hamilton Rating Scale for Depression, 17 items (HDRS-17) | Weeks 0 and 6
  Continuous measure (score changes).

SECONDARY OUTCOMES:
Change in HDRS-17 | Weeks 1, 2, 4, 6, 8, 12
  Continuous measure (score changes).
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Weeks 1, 2, 4, 6, 8, 12
  Continuous measure (score changes).
Change in Global Clinical Impression Scale (CGI) | Weeks 1, 2, 4, 6, 8, 12
  Continuous measure (score changes).
Change in Cumulative Illness Rating Scale (CIRS) | Weeks 1, 2, 4, 6, 8, 12
  Continuous measure (score changes).
Change in Geriatric Depression Scale (GDS) | Weeks 1, 2, 4, 6, 8, 12
  Continuous measure (score changes).
Change in Positive and Negative Affect Scale (PANAS) | Weeks 1, 2, 4, 6, 8, 12
  Continuous measure (score changes).
Change in serum BDNF concentrations | Weeks 0 and 6
  Continuous measure (score changes).
Response HDRS 17 | Week 12
  Response (≥50% improvement from week 0 to 12)
Remission of HDRS 17 | Week 12
  Remission (HDRS-17 ≤ 8)
Young Manic Rating Scale (YMRS) | Weeks 0, 1, 2, 4, 6, 8, 12
  Serious adverse events include treatment-emergent hypomania/mania (YMRS>8), suicide, psychiatric hospitalization and others life-threatening or incapacitant events
Serious adverse events | Up to week 12
  Serious adverse events include treatment-emergent hypomania/mania (YMRS>8), suicide, psychiatric hospitalization and others life-threatening or incapacitant events

OTHER OUTCOMES:
Conditioned pain modulation | Week 0 and 4
  Temperature of the thermode reported as painful
Actigraphy | 1 week before treatment up to 4 weeks after finishing study
  Continuous measure (score changes).

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Valiengo, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Valiengo L, Pinto BS, Marinho KAP, Santos LA, Tort LC, Benatti RG, Teixeira BB, Miranda CS, Cardeal HB, Suen PJC, Loureiro JC, Vaughan RAR, Dini Mattar RAMPF, Lessa M, Oliveira PS, Silva VA, Gattaz WF, Brunoni AR, Forlenza OV. Treatment of depression in the elderly with repetitive transcranial magnetic stimulation using theta-burst stimulation: Study protocol for a randomized, double-blind, controlled trial. Front Hum Neurosci. 2022 Aug 31;16:941981. doi: 10.3389/fnhum.2022.941981. eCollection 2022. PMID 36118977

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT04842929/Prot_SAP_002.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT04842929/ICF_003.pdf